CLINICAL TRIAL: NCT02169973
Title: An Open-Label Study to Investigate the Regional Brain Kinetics of the Positron Emission Tomography Ligand 11C-MK-3168 and the Blocking of the Retention of the Ligand in the Human Brain by JNJ-42165279
Brief Title: A Study to Investigate the Regional Brain Kinetics of the Positron Emission Tomography Ligand 11C-MK-3168 and the Blocking of the Retention of the Ligand in the Human Brain by JNJ-42165279
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR103601; 42165279EDI1003 (Other: Janssen Research & Development, LLC); 2013-004199-37 (EudraCT Number)
Record Dates: First submitted 2014-02-26; First posted 2014-06-23 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Healthy; Positron Emission Tomography; 11C-MK-3168; JNJ-42165279; Human Brain
MeSH Terms: interventions — JNJ-42165279

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A (Experimental): 3 to 5 participants will undergo Positron Emission Tomography (PET)/computed tomography scan after administration of 11C-MK-3168 on Day 1.
  Interventions: Drug: 11C-MK-3168
- Part B (Experimental): 3 to 12 participants will undergo PET scan after administration of 11C-MK-3168 on Day 1. Participants will receive 2 single doses of JNJ-42165279: 100 mg on Days 1 and up to 250 mg on Day 8. Participants will undergo PET scans after 1 hour of each administration of JNJ-42165279 on Days 1 and 8, with 11C-MK-3168 administration.
  Interventions: Drug: JNJ-42165279; Drug: 11C-MK-3168
- Part C (Experimental): 4 to 8 participants will undergo PET scan after administration of 11C-MK-3168 on Day 1. Participants will receive once daily dose of JNJ-42165279 (up to 100 mg) from Day 1 to Day 7. Participants will undergo PET scans after 24 hour of administration of JNJ-42165279 on Days 1 and 7, with 11C-MK-3168 administration.
  Interventions: Drug: JNJ-42165279; Drug: 11C-MK-3168

INTERVENTIONS:
Drug: JNJ-42165279 — Participants will receive oral suspension of JNJ-42165279 in Part B as single dose on Day 1 (100 mg) and on Day 8 (up to 250 mg); in Part C as once daily dose (up to 100 mg) from Day 1 to Day 7.
  Arms: Part B; Part C
Drug: 11C-MK-3168 — Participants will receive 11C-MK-3168 in the target range of 185 to 370 megabecquerel (MBq) intravenously (into a vein) before every positron emission tomography scan in Parts A, B, and C.

SUMMARY:
The purpose of the study is to measure the uptake, distribution, and clearance of 11C-MK-3168 by Positron Emission Tomography (PET) scan and to model the tissue specific kinetics of 11C-MK-3168 with the appropriate input function in human brain in Part A; to measure blocking of retention of 11C-MK-3168 at the estimated time to maximum plasma concentration after dosing (tmax) following each single oral doses of JNJ-42165279 and model the exposure/enzyme interaction of JNJ-42165279 in Part B; to measure the saturation of enzyme inhibition in the brain at steady state plasma concentrations of JNJ-42165279 (on Day 8) after 7 once-daily doses of JNJ-42165279 by conducting PET studies with 11C-MK-3168 at trough plasma concentrations on Day 2 in Part C.

DETAILED DESCRIPTION:
This is an open-label (both [participants and investigator] know what treatment participants will receive) study. This study consists of 3 consecutive parts: A, B, and C. Each part will consist of a screening phase (between 21 to 2 days prior to the study medication), a treatment phase (Part A: 1 day; Part B: 8 days; Part C: 8 days), and the end-of-study/ follow-up visit (within 5 to 7 days after last PET scan). In the treatment phase of the Part A, participants will undergo a baseline PET/computed tomography scan (after administration of 11C-MK-3168 on Day 1); In Part B, participants will undergo a baseline PET scan, followed by 2 post-treatment PET scans after 2 single doses of JNJ-42165279 on Days 1 and 8; in Part C, participants will undergo a baseline PET scan, followed by 2 post-treatment PET scans after 24 hours postdose of JNJ-42165279 on Days 1 and 7. Safety will be evaluated by the assessment of adverse events, vital signs, 12-lead electrocardiogram, clinical laboratory testing, physical examination (including weight and tympanic temperature [temperature measure in an ear]), and neurological examination. The total duration of study participation for a participant will be approximately 4 weeks for Part A and approximately 5 weeks for Parts B and C.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 30 kg/m2 inclusive (BMI = weight/height2)
* Non-smoker (not smoked for 3 months prior to screening)
* Agree to use one of the protocol mentioned barrier methods of birth control

Exclusion Criteria:

* Exposed to 1 millisievert or more of ionizing radiation in the year before the start of this study
* Clinically significant abnormal laboratory values and abnormal physical and neurological examination at screening
* Any clinically significant Magnetic Resonance Imaging (MRI) abnormalities at screening, as determined by a neuroradiologist, which are relevant for the study
* Allen test (test to assess the arterial blood flow to the hand) indicating abnormal blood supply to the hand
* Has implanted or embedded metal objects, or fragments in the head or body that would present a risk during the MRI scanning procedure

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Part A: Compartmental Model of the Volume of Distribution of 11C-MK-3168 in Brain by Positron Emission Tomography (PET) | Day 1
  Uptake, distribution, and clearance of 11C-MK-3168 in the brain and plasma of healthy male participants will be evaluated by PET scan and arterial sampling.
Part B: Dose Dependent Occupancy of Fatty Acid Amide Hydrolase (FAAH) After Single Dose of JNJ-42165279 | Up to 5 weeks
  Occupancy of the FAAH in brain by JNJ-42165279 will be evaluated by comparing the distribution volume of 11C-MK-3168 after single dose JNJ-42165279 to the distribution volume at baseline.
Part C: Dose and Time Dependent Occupancy of FAAH After Repeat Dose of JNJ-42165279 | Upto 5 weeks
  Occupancy of FAAH in brain by JNJ-42165279 at steady state will be evaluated by comparing the distribution volume of 11C-MK-3168 at Tmax after single dose JNJ-42165279 and then at trough after dosing for seven days with JNJ-42165279 to the distribution volume prior to treatment.

SECONDARY OUTCOMES:
Correlation Between Fatty Acid Amide Hydrolase (FAAH) Occupancy in Brain With Peripheral FAAH inhibition | Postdose Day 1 and Day 8
  Correlation between peripheral and central FAAH inhibitions in white blood cells by JNJ 42165279 will be measured.
Effect of FAAH C385A polymorphism on the distribution volume of 11C-MK-3168 in human brain | Postdose Day 1 and Day 8
  Effect of FAAH C385A polymorphism on the distribution volume of 11C-MK-3168 in human brain will be assessed.
Number of participants with adverse events | Up to 5 weeks
  Number of participants with adverse events will be reported as an assessment of safety and tolerability of 11C-MK-3168 and JNJ-42165279.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Leuven, Belgium